CLINICAL TRIAL: NCT07205484
Title: Early Communication Intervention for Deaf/Hard of Hearing Toddlers: Long-Term Language and Literacy Outcomes
Brief Title: Long-Term Outcomes of Early Communication Intervention for Deaf/Hard of Hearing Toddlers
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R01DC016877-06A1 (NIH)
Record Dates: First submitted 2025-08-06; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Bilateral
Keywords: Hearing Loss; School-Aged Outcomes; Language; Literacy; Early Intervention; Parent-Mediated Intervention
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss; Language; Literacy

STUDY DESIGN:
Intervention Model Description: Parent-child dyads were randomly assigned to the parent-mediated intervention (PMI) or business-as-usual (BAU) control group. Randomization was stratified on hearing device and communication mode. Hearing device was dichotomized as either (1) hearing aid or (2) cochlear implant, cochlear implant candidate, or bone conduction device. Communication mode was dichotomized as using visual communication with the child (1) less than 10% of the time or (2) 10% or more of the time.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and coders will be naive to the experimental condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-Mediated Intervention (PMI) (Experimental): Participants in both the parent-mediated intervention (PMI) group and the business-as-usual (BAU) control group continued to receive standard community-based early intervention services outside of the clinical trial. In addition to these services, dyads in the PMI group participated in weekly intervention sessions via Zoom for 6 months.
  Intervention sessions followed a Teach-Model-Coach-Review framework to support parents in using communication support strategies with their child. Parents were taught seven communication support strategies in a fixed sequence: (1) Setting the Stage, (2) Play and Engage, (3) Respond and Wait, (4) Notice and Say, (5) Show It, (6) Contrast It, and (7) Add On. These strategies focused on helping parents create opportunities for language learning during everyday routines and play, notice and respond to their child's communication, and model rich, salient language.
  Interventions: Behavioral: Parent-Mediated Intervention (PMI)
- Business-As-Usual (BAU) Control (No Intervention): Participants in both the parent-mediated intervention (PMI) group and the business-as-usual (BAU) control group continued to receive standard community-based early intervention services outside of the clinical trial. Dyads in the BAU control group did not receive the PMI.

INTERVENTIONS:
Behavioral: Parent-Mediated Intervention (PMI) — The PMI consisted of weekly, 1-hour intervention sessions via Zoom for 6 months. In total, the intervention consisted of 26 intervention sessions.
  Other Names: Parent-Implemented Communication Intervention (PICT); Parent-Implemented Communication Treatment (PICT)
  Arms: Parent-Mediated Intervention (PMI)

SUMMARY:
The overall goal of this randomized clinical trial is to learn about the effects of a parent-mediated intervention (PMI) designed to support communication outcomes for deaf and hard-of-hearing (DHH) children. Previously, the investigators enrolled 96 DHH children between 12 and 18 months of age and their parents. Families were randomly assigned to receive either the PMI or a business-as-usual control group. The PMI was a 6-month intervention that included weekly, hour-long Zoom sessions. During the intervention sessions, parents were taught communication support strategies to support their child's language development throughout daily routines and play.

This current period of the trial follows the same children into early elementary school to determine whether the effects of the PMI are long-lasting. The main questions it aims to answer are:

* Does the PMI improve language, reading, and social communication outcomes in the early school years?
* Does parent involvement during early intervention support continued engagement in their child's education?

The investigators will compare parents and children who received the PMI to those in the business-as-usual control group to determine whether the intervention has lasting effects on these outcomes.

Participants will complete standardized assessments, parent-report surveys, and video-recorded naturalistic interactions. All assessments will be completed remotely.

DETAILED DESCRIPTION:
Hearing loss is one of the most prevalent congenital conditions. Recent advances in early detection and technology have contributed to significant improvements in long-term outcomes for deaf/hard-of-hearing (DHH) children. Despite this progress, language and literacy outcomes for school-age DHH children are inconsistent, and many DHH children do not "catch up" to their hearing peers. Closing this gap requires the implementation of effective early communication interventions. Yet, until recently, there was a significant paucity of research on early communication interventions for DHH children. Parent-mediated interventions (PMIs), which involve teaching parents strategies to enhance their child's language learning experiences, are a promising form of early intervention for DHH toddlers. During the previous project period (NCT03803943), 96 DHH children, between 12 and 18 months of age and their parents, were enrolled. Parent-child dyads were randomly assigned to receive either the PMI or business-as-usual control group. The investigators examined the effects of the intervention on (a) parent strategy use and (b) child communication outcomes during and after the 6-month intervention period. The follow-up period of the clinical trial is outlined here.

This trial will be the first large-scale evaluation of the long-term effects of an early communication intervention on school-age language and literacy outcomes for DHH children. The study enrolled 96 parent-child dyads, 88 of whom remain involved and consented to contact for the follow-up period. The investigators will complete follow-up assessments during early elementary school. The investigators plan to examine the long-term effects of the intervention on school-age outcomes and characterize the intermediary mechanisms of these effects. The investigators consider not only how early communication interventions affect subsequent child outcomes, but also how involving parents early in their child's development may lay the foundation for sustained parent engagement as children transition to school-based services. Taken together, the investigators plan to integrate child and parent outcomes to fully characterize how early language learning experiences shape long-term language and literacy outcomes. Understanding the pathways through which early interventions affect the developmental trajectory of DHH children will have widespread implications for research and clinical practice.

ELIGIBILITY:
Eligibility for the follow-up period of the clinical trial is dependent on enrollment in the initial period of the clinical trial.

Child inclusion criteria were:

* between 12-18 months
* diagnosed with bilateral hearing loss
* no additional diagnoses (e.g., Down syndrome, cerebral palsy, seizure disorder, blindness, etc.)
* one parent with typical hearing
* exposed to some degree of spoken language by their parents.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Evaluation of Language Fundamentals, Fifth Edition (CELF-5) | 7 - 8 years old
  The Clinical Evaluation of Language Fundamentals, Fifth Edition (CELF-5) is a standardized assessment of language development. The Core Language Standard Score (M = 100, SD = 15) reflects the child's global language ability, with higher scores indicating better language skills.
Peer-Peer Interaction, Pragmatic Observational Measure (POM) | 7 - 8 years old
  The Pragmatic Observational Measure (POM), a rating scale of pragmatic skills, will be scored during a naturalistic peer-peer interaction. The POM includes 27 items, capturing a range of pragmatic skills, rated on a 4-point scale (1 = rarely or never observed; 4 = almost always observed). The POM Total Raw Score (Min = 27, Max = 108) reflects the child's pragmatic skills, with higher scores indicating better pragmatic skills.
Woodcock Reading Mastery Tests, Third Edition (WRMT-III) | 7 - 8 years old
  The Woodcock Reading Mastery Tests, Third Edition (WRMT-III) is a standardized assessment of reading development. The Total Reading Cluster Standard Score (M = 100, SD = 15) reflects the child's global reading ability, with higher scores indicating better reading skills.

SECONDARY OUTCOMES:
Parent-Child Interaction, Keys to Interactive Parenting Scale (KIPS) | 5 - 6 years old
  The Keys to Interactive Parenting Scale (KIPS), a rating scale of parenting behaviors, will be scored during a naturalistic parent-child interaction.The KIPS includes 12 items, capturing a range of parenting behaviors, rated on a 5-point scale, with higher scores reflecting higher quality parent behaviors. The KIPS Total Mean Score (Min = 1.0, Max = 5.0), calculated as the average of all 12 items, reflects the overall quality of parenting behaviors.
Parent Empowerment and Efficacy Measure (PEEM) | 5 - 6 years old
  The Parent Empowerment and Efficacy Measure (PEEM) is a self-report questionnaire assessing parents' confidence in their role and their ability to support their child's development. The measure includes 20 items rated on a 10-point scale (1 = no agreement; 10 = complete agreement). The PEEM Total Raw Score (Min = 20, Max = 200) reflects overall parenting self-efficacy, with higher scores indicating greater self-efficacy.
Parental Involvement Survey in Their Child's Elementary Studies (PISCES) | 5 - 6 years old
  The Parental Involvement Survey in Their Child's Elementary Studies (PISCES) is a parent-report questionnaire that assesses parent involvement in school-related activities. The measure includes 56 items rated on a 4-point Likert scale (1 = strongly disagree; 4 = strongly agree). The PISCES Total Raw Score (Min = 56, Max = 224) reflects the extent of parent involvement in their child's education, with higher scores indicating greater involvement.
The Parent Advocacy Skills and Comfort Survey | 5 - 6 years old
  The Parent Advocacy Skills and Comfort Survey is a parent-report questionnaire assessing caregivers' ability to advocate for their child's educational needs. The survey includes 10 items rated on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree). The Total Raw Score (Min = 10, Max = 50) reflects overall advocacy skills and confidence, with higher scores indicating greater advocacy skills and confidence.
Clinical Evaluation of Language Fundamentals, Fifth Edition (CELF-5) | 5 - 6 years old
  The Clinical Evaluation of Language Fundamentals, Fifth Edition (CELF-5) is a standardized assessment of language development. The Core Language Standard Score (M = 100, SD = 15) reflects the child's global language ability, with higher scores indicating better language skills.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, CCC-SLP, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All participant-level data related to the primary and secondary outcomes of the clinical trial will be preserved and shared via Dryad. All shared data will be de-identified by using a unique study identifier and age in months rather than date of birth. This will allow for the replication of all analyses for the primary aims and for other investigators to answer other questions that are not related to the study aims. The final results of the study will be uploaded to clinicaltrials.gov.
  All data as described above will be shared, as allowed by informed consents. The only data that will not be shared are the video recordings of the observational peer-peer and parent-child interactions, which contain participants' faces.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available no later than the time of publication of the main study aims or the end of the project period, whichever comes first. Data will be stored and available via Dyrad in perpetuity.
Access Criteria: Dryad datasets are indexed by the Thomas-Reuters Data Citation Index, Scopus, and Google Dataset Search. Dyrad gives each dataset a unique Digital Object Identifier, which when entered into any browser will take the user to the landing page of the dataset.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT07205484/ICF_000.pdf